CLINICAL TRIAL: NCT00925275
Title: A Phase I, Multi-Center, Open-Label, Dosimetry Study of I-131-CLR1404 in Patients With Relapsed or Refractory Advanced Solid Tumors Who Have Failed Standard Therapy or for Whom No Standard Therapy Exists
Brief Title: Dosimetry Study of I-131-CLR1404 in Patients With Relapsed or Refractory Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar, Inc (Industry)
Responsible Party: Director Clinical Operations, Cellectar, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DCL-08-001
Record Dates: First submitted 2009-06-18; First posted 2009-06-22 (Estimated); Last update posted 2010-05-04 (Estimated); Status verified 2010-04

CONDITIONS: Solid Tumors
Keywords: Solid tumors; Refractory; Relapsed; Radiation; Dosimetry; Radiopharmaceutical; Biodistribution; Pharmacokinetics; Cancer; Phase I
MeSH Terms: conditions — Recurrence; Neoplasms | interventions — CLR1404; lortalamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dosimetric (Experimental)
  Interventions: Drug: I-131-CLR1404

INTERVENTIONS:
Drug: I-131-CLR1404 — Single intravenous injection of 10 millicuries of I-131-CLR1404 given on Day 0
  Other Names: CLR1404; 1404

SUMMARY:
The purpose of the study is to investigate the safety, biodistribution, radiation dosimetry and pharmacokinetics of I-131-CLR1404.

DETAILED DESCRIPTION:
I-131-CLR1404 is a small-molecule, phospholipid ether analog that combines lipid-like properties with a cancer therapeutic beta-emitting radioisotope. Cellectar believes that this compound will benefit individuals with cancer due to its selective retention and accumulation in malignant cells versus nonmalignant cells. Preclinical experiments have demonstrated that I-131-CLR1404 significantly slows malignant tumor growth in several mouse tumor models.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory advanced solid tumor(s) and have exhausted standard treatment options or no standard therapy exists
* Must have a sufficient window of time to complete the washout period, dosimetry data acquisition and the follow up safety assessment period
* ECOG performance status of 0 or 1 and estimated life expectancy of ≥ 4 months
* 18 years or older
* Must be compliant with the protocol and be within geographical proximity to make the required study visits
* Have the ability to read, understand and provide written informed consent
* Patients with brain metastasis are acceptable if the clinical condition has been stable for at least one month
* Female patients of childbearing potential must have a negative serum pregnancy test within 24 hours of start of treatment
* Must agree to use an effective method of contraception during the study and for 90 days following the last dose of study drug

Exclusion Criteria:

* Patient or physician plans concomitant chemotherapy, therapeutic radiation treatment, and/or biological treatment for cancer including immunotherapy while on study
* More than 25% of the total bone marrow irradiated
* Diffuse lung disease or interstitial spread of carcinoma
* Bladder or rectum is within a prior radiation therapy field and a dose of greater than 45 Gy was administered
* Total therapeutic radiation dose in the past year in excess of 25 Gy to the kidney, 45 Gy to brain, 45 Gy to stomach, 18 Gy to lung, or 25 Gy to liver
* Prior total-body irradiation
* Extradural tumor in contact with the spinal cord, or tumor located where swelling in response to therapy may impinge upon the spinal cord
* Prior radiation therapy or chemotherapy within 2 weeks of the start of the study
* Active medical condition(s) or organ disease(s) that may either compromise patient safety or interfere with the safety and/or outcome evaluation of the study drug
* Laboratory values ≤ 7 days:

  * WBC < 3000/µL
  * Absolute neutrophil count < 1500/µL
  * Platelets < 150,000/µL
  * Hemoglobin ≤ 11.0 gm/dL
  * Total bilirubin > 1.5 x upper limit of normal for age
  * SGOT or SGPT > 3 x upper limit of normal for age if no liver metastases or > 5 x upper limit of normal for age in the presence of liver metastases
  * Serum creatinine > 1.5 x upper limit of normal for age
  * INR ≥ 2.0
* Investigational drug, investigational biologic, or investigational therapeutic device within 30 days of initiating study drug
* Severely marrow toxic drugs (e.g. nitrosoureas, mitomycin)
* Prior treatment with Iodine-131 in the past five years
* Concurrent hemodialysis
* Blood transfusions within 60 days of study start
* Hematopoietic growth factor therapy within 60 days of study start
* Prior stem cell transplantation
* Clinically evident ascites or with peritoneal carcinomatosis
* Clinically significant cardiac co-morbidities including: CHF, a LVEF< 40%, unstable angina pectoris, serious cardiac arrhythmia requiring medication or a pacemaker, myocardial infarction within the past six months
* Clinically significant pulmonary impairment defined as an SaO2 on room air of 93% or less
* Concurrent or recent use of thrombolytic agents, or full-dose anticoagulants
* Uncontrolled hypertension or patients with uncontrolled diabetes
* Grade II-IV peripheral vascular disease or peripheral vascular surgery within the past year
* Less than 4 weeks since prior major surgery
* Known positive for HIV, Hepatitis C (active, previously treated or both), or is Hepatitis B core antigen positive
* Concurrent chronic use of aspirin (325 mg/day or more)
* Pregnant or lactating
* Patients with colostomy/ileostomy
* Poor venous access
* Prior allergic reactions to iodine, or other study agents
* Significant traumatic injury within the past 4 weeks
* Ongoing or active infection requiring antibiotics or with a fever >38.1°C (>101° F) within 3 days of the first scheduled day of dosing
* Patients who are hospitalized

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Calculate whole body and organ radiation dosimetry of I-131-CLR1404 to determine the millicurie dose which is expected to deliver 35-40 centigray of radiation to bone marrow | 42 days

SECONDARY OUTCOMES:
To determine the safety and pharmacokinetic profile of I-131-CLR1404 | 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Cellectar, Inc
Locations (4):
- United States (4):
  - City of Hope, Duarte, California
  - Georgetown University, Lombardi Cancer Center, Washington D.C., District of Columbia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Grudzinski JJ, Titz B, Kozak K, Clarke W, Allen E, Trembath L, Stabin M, Marshall J, Cho SY, Wong TZ, Mortimer J, Weichert JP. A phase 1 study of 131I-CLR1404 in patients with relapsed or refractory advanced solid tumors: dosimetry, biodistribution, pharmacokinetics, and safety. PLoS One. 2014 Nov 17;9(11):e111652. doi: 10.1371/journal.pone.0111652. eCollection 2014. PMID 25402488